CLINICAL TRIAL: NCT05391841
Title: Prospective, Non-interventional Study to Evaluate the Efficacy and Safety of NOVOCART Inject for the Treatment of Cartilage Defects in the Knee in Pediatric Patients With Closed Epiphyses
Brief Title: Non-interventional Study in Pediatric Patients Treated With NOVOCART Inject in the Knee
Acronym: NINJA
Status: Withdrawn | Type: Observational
Why Stopped: A waiver was granted for paediatric patients. Therefore, the study is not necessary.
Sponsor: Tetec AG (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2123
Record Dates: First submitted 2022-04-08; First posted 2022-05-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-05

CONDITIONS: Cartilage Disease
Keywords: NOVOCART Inject; Cartilage Defect; Pediatric Patients; Knee; Cartilage Injury
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: NOVOCART Inject — Autologous Chondrocyte Implantation

SUMMARY:
The study is a prospective, multicenter, single-arm non-interventional study to evaluate the efficacy, safety and health economics of NOVOCART® Inject in the treatment of cartilage defects of the knee in pediatric patients with radiologically proven closed epiphyseal growth plates.

DETAILED DESCRIPTION:
In this non-interventional study NOVOCART® Inject, which is marketed in Germany under a license according to Section 4b of the AMG, will be used in routine clinical practice according to the current authorized Summary of Product Characteristics (SmPC). As stated in this SmPC, NOVOCART® Inject may only be used by physicians who are trained on the product. The treatment with NOVOCART® Inject requires two surgeries. During the first surgery cartilage tissue will be harvested arthroscopically and sent to TETEC AG for NOVOCART® Inject manufacturing, then NOVOCART® Inject will be transplanted during a second surgery about 3 to 4 weeks later.

All patients will be followed up for 5 years post NOVOCART® Inject implantation and data will be collected preoperatively and at 3, 6, 12, 18, 24, 36, 48 and 60 months as outlined at the end of this synopsis.

NOVOCART® Inject post treatment rehabilitation should follow the recommendations given in the SmPC and during product training.

The primary and secondary variables (see below) will be assessed after a follow-up of 24 month post NOVOCART® Inject implantation (primary analysis).

Long-term data will be assessed after an additional 3 years follow-up (follow-up analysis).

The collected data will be documented using dedicated case report forms (CRFs) which are created by TETEC AG.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (< 18 years of age at implantation)
* Closure of the epiphysis adjacent to the biopsy harvest site or the defect to be treated confirmed by an adequate imaging modality
* Localized full-thickness cartilage defect (ICRS grade III or IV) of the knee
* Medicinal indication for NOVOCART® Inject treatment

Exclusion Criteria:

see NOVOCART Inject SmPC

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (< 18 years of age) with closed epiphyses who suffer from a full-thickness cartilage defect of the knee caused by acute or repetitive trauma or by osteochondrosis dissecans and who are scheduled for treatment with NOVOCART Inject SmPC, where the therapeutic indications, contraindications, special warnings and precautions for use are listed in detail. The decision to treat patients with NOVOCART Inject must be made independently from the patient's participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Responder rate of overall KOOS | 24-months Follow-up
  The overall Knee injury and Osteoarthritis Outcome Score (KOOS5) responder rate defined as the proportion of patients with ≥ 10 points improvement in the KOOS5 from baseline.

SECONDARY OUTCOMES:
Change of overall KOOS from baseline | 24-months Follow-up
  Change of overall KOOS from baseline to the 24-month assessment, Knee Injury and Osteoarthritis Outcome Score, score 0-100, higher score shows better outcome
Change of the 5 sub-scores of the KOOS from baseline | 24-months Follow-up
  Change of the 5 sub-scores of the KOOS from baseline to the 24-month assessment, Knee Injury and Osteoarthritis Outcome Score, score 0-100, higher score shows better outcome
Change of the IKDC subjective score from baseline | 24-months Follow-up
  Change from baseline to the 24-month visit in the IKDC subjective score, international knee documentation committee, score 0-100, higher score shows better outcome
Change in the IKDC surgeon's part from baseline | 24-months Follow-up
  Change from baseline to the 24-month visit in the IKDC surgeon's part. international knee documentation committee, score 0-100, higher score shows better outcome
MOCART (MRI imaging) | 24-months Follow-up
  In vivo performance measured by the assessment of the Magnetic Resonance, Observation of Cartilage Repair Tissue (MOCART) score, Magnetic Resonance Observation of Cartilage Repair Tissue, score 0-100, higher score shows better outcome
IKDC subjective score responder rate | 24-months Follow-up
  IKDC subjective score responder rate, defined as the proportion of patients with > 20.5 points improvement in the IKDC subjective score from baseline to the 24-month visit
Proportion of patients with treatment failure | 24-months Follow up, 60-months Follow-up
  Proportion of patients with treatment failure
Number of postop physical therapy | 24-months Follow up, 60-months Follow-up
  Number of postop physical therapy
Number of postop doctor visits | 24-months Follow up, 60-months Follow-up
  Number of postop doctor visits
Days of hospitalisation | 24-months Follow up, 60-months Follow-up
  Days of hospitalisation
Work/school status checklist | 24-months Follow up, 60-months Follow-up
  Work/school status, changes due to injury in work or school status (pupil, worker full or part time, not working, job seeking)
Days of work/school missed | 24-months Follow up, 60-months Follow-up
  Days of work/school missed
Patient satisfaction | 24-months Follow up, 60-months Follow-up
  Patient questionnaire, 4 questions with 3 answer choices better, same, worse
Treatment-related adverse reactions (ARs) | 24-months Follow up, 60-months Follow-up
  Treatment-related adverse reactions (ARs)
Rate of unplanned re-operations | 24-months Follow up, 60-months Follow-up
  Rate of unplanned re-operations: all unplanned reoperations and those related to NOVOCART® Inject treatment
Surgical time | 24-months Follow up, 60-months Follow-up
  cut-to-suture time
Length of incision | 24-months Follow up, 60-months Follow-up
  Length of incision

OTHER OUTCOMES:
Adverse reactions | 24-months Follow up, 60-months Follow-up
  Continuous assessment of adverse reactions (ARs)
Number of device deficiencies - trephine | 24-months Follow up, 60-months Follow-up
  Number of device deficiencies - trephine
Number of device deficiencies - Application System | 24-months Follow up, 60-months Follow-up
  Number of device deficiencies - Application System
Number of device deficiencies - number of product related issues | 24-months Follow up, 60-months Follow-up
  Number of device deficiencies - number of product related issues

CONTACTS AND LOCATIONS:
Overall Officials: Peter Angele, Prof. Dr., Principal Investigator — Universitätsklinik Regensburg
Locations (6):
- Germany (6):
  - St. Josefs-Hospital Cloppenburg gemeinnützige GmbH, Cloppenburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - OCM Klinik GmbH München, München
  - Klinikum rechts der Isar, Technische Universität München, München
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No